CLINICAL TRIAL: NCT03905161
Title: Does Rhythmic Auditory Stimulation Influence Walking Speed in the 6-minute Walk Test in Patients With Myasthenia Gravis?
Brief Title: Rhythmic Auditory Stimulation and Walking Speed in the 6-minute Walk Test
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Linda Kahr Andersen, Research Physiotherapist, PhD student, Rigshospitalet, Denmark
Other Study IDs: H-18031231 3
Record Dates: First submitted 2019-04-02; First posted 2019-04-05 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Myasthenia Gravis
Keywords: Fatigue; 6-minute walk test; Rhythmic Auditory Stimulation
MeSH Terms: conditions — Myasthenia Gravis; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myasthenia patients: Danish patients with myasthenia gravis seen at the Department of Neurology, Rigshospitalet
  Interventions: Other: 6-minute walk test

INTERVENTIONS:
Other: 6-minute walk test — The 6-minute walk test (6MWT) is widely used in the clinic to measure treatment efficacy and disease progression in patients with neuromuscular diseases and is found valid and reliable to measure decrease in walking speed for neuromuscular patients.

SUMMARY:
The aim of this study is to investigate if rhythmic auditory stimulation can influence walking speed, during a 6MWT in patients with myasthenia gravis (MG).

DETAILED DESCRIPTION:
Background

1. The 6-minute walk test (6MWT) is widely used in the clinic to measure treatment efficacy and disease progression in patients with neuromuscular diseases and is found valid and reliable to measure decrease in walking speed.
2. Rhythmic auditory stimulation has repeatedly been shown to improve gait parameters in individuals with neurologic impairment.

The aim of this study is to investigate if rhythmic auditory stimulation can influence walking speed, during a 6MWT in patients with myasthenia gravis.

Patients with MG are asked to complete two 6MWTs separated by minimum 30 minutes of rest. Before the 6MWTs patient is instructed to walk 60 m as fast as possible, and their steps per minute (SPM) is recorded. When completing the 6MWTs, one of the tests is accompanied by music (m6MWT) with a beat per minute (BPM) corresponding to patients' SPM. The order of the 6MWTs is randomly decided by pre-ordered sealed envelopes.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed informed consent.
* Able to read and understand Danish or English.
* Diagnosis of mild to moderate MG (Able to provide signed informed consent.

  * Able to read and understand Danish or English.
  * Diagnosed with generalized mild to moderate myasthenia gravis (I-IV on the Myasthenia Gravis Foundation of American Clinical Classification, MGFA).
  * Documented history of acetylcholine receptor (AChR) or Muscle Specific Kinase (MuSK) antibody positive, or abnormal repetitive nerve stimulation testing (decrement > 10%) on electromyography (EMG) or abnormal single fiber EMG (conduction block or jitter) or based on their clinical history and symptom improvement with acetylcholinesterase inhibitors.
* Ability to walk > 60 meters in a 6MWT.

Exclusion Criteria:

MGFA grade V disease

* Other disorders that are not related to MG, or drugs, that interfere with muscle strength, walking ability, balance and fatigue (e.g. heart failure).
* Serious medical illness (e.g. uncontrolled insulin dependent diabetes mellitus, symptomatic coronary artery disease, and cancer).
* Dementia or pregnancy.
* Unspecified reasons judged by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MG seen in the Department of Neurology, Rigshospitalet, fulfilling the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
6-minute walk test (6MWT) | 6 minutes
  The distance (meter) and walking speed (meter per seconds) in a 6-minute walk test.

SECONDARY OUTCOMES:
Heart rate | 5 minutes
  Monitoring of heart rate by a pulse-watch prior, during (average heart rate for 6 minutes) and after the 6MWT. All three measurements are in the same units (beats per minute), and are registered directly from the pulse-watch, which the patient wear during the walk test.
The Borg Rating of Perceived Exertion (RPE) scale. | 2 minutes
  Just after the completed 6MWT patients are asked to score the perceived exertion during walking. The scale is from 6 (no effort at all) to 20 (absolute maximal effort).
Myasthenia gravis composite score (MGC) | 30 minutes
  The Myasthenia Gravis composite score (MGC) covers 10 important functional domains most frequently involved in patients with MG. This scoring system is based on quantitative testing of muscle groups, or symptom history told by the patient, by means of a 4 point scale ranging from 0 (no symptoms) to 9 (severe symptoms). The scale measures ocular, bulbar, respiratory and limb function, grading each finding, and the total score ranges from 0(no myasthenic findings) to 50 (maximal myasthenic deficits).

CONTACTS AND LOCATIONS:
Overall Officials: Linda K Andersen, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark